CLINICAL TRIAL: NCT05146882
Title: A Phase 2 Open-Label Extension Study to Evaluate the Safety and Pharmacodynamics of Belcesiran in Patients With PiZZ Alpha-1 Antitrypsin Deficiency Associated Liver Disease
Brief Title: An Extension Study of Belcesiran in Patients With Alpha-1 Antitrypsin Deficiency Associated Liver Disease (AATLD)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Update to Program Design - No Participants Enrolled
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DCR-A1AT-202; STARLIGHT (Other: Dicerna Pharmaceuticals)
Record Dates: First submitted 2021-11-09; First posted 2021-12-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- belcesiran (Experimental): Participants who completed the DCR-A1AT-201 treatment period will receive open-label belcesiran administered subcutaneously
  Interventions: Drug: Belcesiran
- Observational (No Intervention): Participants who completed the DCR-A1AT-201 Conditional Follow-up period will enter DCR-A1AT-202 for continued follow-up (will not receive open-label belcesiran)

INTERVENTIONS:
Drug: Belcesiran — Belcesiran will be administered subcutaneously (SC) in the treatment arm.
  Arms: belcesiran

SUMMARY:
This is a Phase 2, multicenter, open-label extension of Study DCR-A1AT-201, designed to evaluate the long-term safety and further characterize the pharmacodynamics (PD) of belcesiran in adult patients with PiZZ AATLD.

ELIGIBILITY:
Inclusion Criteria:

1. Must be 18 to 75 years of age inclusive, at the time of signing the Informed Consent Form (ICF).
2. Documented diagnosis of PiZZ-type Alpha-1 Antitrypsin deficiency (AATD), confirmed by genotyping.
3. Lung, renal and liver function within acceptable limits.
4. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

1. Any condition that, in the opinion of the Investigator, would make the participant unsuitable for enrollment or could interfere with participation in or completion of the study
2. Routine use of acetaminophen/paracetamol
3. Use of systemically acting steroids in the month prior to Screening and throughout the study period.
4. Positive SARS-CoV-2 virus test at Screening
5. Any other safety laboratory test result considered clinically significant and unacceptable by the Investigator
6. Inability or unwillingness to comply with the specified study procedures, including lifestyle considerations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
The incidence of treatment-emergent adverse events | up to 152 weeks
The change from baseline in pulmonary function tests (PFTs) | up to 152 weeks
  Forced expiratory volume in 1 second (FEV1)
The change from baseline in PFTs | up to 152 weeks
  Forced vital capacity (FVC)
The change from baseline in PFTs | up to 152 weeks
  FEV1/FVC
The change from baseline in PFTs | up to 152 weeks
  diffusing capacity for carbon monoxide (DLCO)
The change from baseline in 12-lead electrocardiogram (ECG) | up to 56 weeks
  heart rate
The change from baseline in ECG | up to 56 weeks
  ventricular rate
The change from baseline in 12-lead ECG | up to 56 weeks
  RR interval
The change from baseline in 12-lead ECG | up to 56 weeks
  PR interval
The change from baseline in 12-lead ECG | up to 56 weeks
  QRS duration
The change from baseline in 12-lead ECG | up to 56 weeks
  QT interval
The change from baseline in 12-lead ECG | up to 56 weeks
  corrected QT interval (QTcF, Fridericia correction)
The change from baseline in physical examination (PE) findings | up to 56 weeks
  body weight
The change from baseline in PE findings | up to 56 weeks
  body-mass index (BMI) (using height from DCR-A1AT-201 study)
The change from baseline in PE findings | up to 56 weeks
  physical examination to assess skin, lungs, cardiovascular system, and abdomen (liver and spleen) based on the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE; version 5.0) grading scale
The change from baseline in vital sign measurements | up to 56 weeks
  blood pressure
The change from baseline in vital sign measurements | up to 56 weeks
  pulse rate
The change from baseline in vital sign measurements | up to 56 weeks
  respiratory rate
The change from baseline in vital sign measurements | up to 56 weeks
  oral temperature
The change from baseline in clinical laboratory tests: Hematology | up to 152 weeks
  Hematology is collected to evaluate the long-term safety of belcesiran
The change from baseline in clinical laboratory tests: Clinical Chemistry | up to 152 weeks
  Clinical Chemistry is collected to evaluate the long-term safety of belcesiran
The change from baseline in clinical laboratory tests: Coagulation | up to 152 weeks
  Coagulation is collected to evaluate the long-term safety of belcesiran
The change from baseline in clinical laboratory tests: Urinalysis | up to 152 weeks
  Urinalysis is collected to evaluate the long-term safety of belcesiran

SECONDARY OUTCOMES:
Changes in serum AAT protein concentrations over time | up to 152 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie Sejling, MD, Study Director — Dicerna Pharmaceuticals
Locations (1):
- Auckland Clinical Studies, Grafton, Auckland, New Zealand